CLINICAL TRIAL: NCT02506465
Title: Multi-center Prospective Study to Assess the Safety and Effectiveness of Medi-Tate i-Temporary Implantable Nitinol Device (iTind) in Subjects With Symptomatic Benign Prostatic Hyperplasia (BPH)
Brief Title: Pivotal Study to Assess the Safety and Effectiveness of the iTind Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medi-Tate Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MT-03
Record Dates: First submitted 2015-07-14; First posted 2015-07-23 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iTind arm (Experimental): iTind implant is implant during the study for 5-7 days.
  Interventions: Device: iTIND
- Sham arm (Sham Comparator): Foley catheter is used during the study
  Interventions: Procedure: Sham Arm

INTERVENTIONS:
Device: iTIND — Temporary Implantable Nitinol Device (iTIND)
  Arms: iTind arm
Procedure: Sham Arm — Foley catheter will be placed and immediately removed.
  Arms: Sham arm

SUMMARY:
The study objectives are to demonstrate the efficacy and safety of the Medi-Tate iTIND as compared to control group (catheter only).

DETAILED DESCRIPTION:
Medi-Tate i-Temporary Implantable Nitinol Device (iTind) is intended to treat subjects with symptomatic BPH.

A total of 150 subjects with symptomatic BPH will be enrolled into this study, according to eligibility criteria.

Study duration is 12 months and includes 7 visits: screening, screening follow up, implantation, retrieval, 6 weeks follow up, 3 months follow up and 12 months follow up.

iTind Device will be implanted for 5-7 days. Sham will be a routine Foley catheter procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signed informed consent form (ICF)
2. Age 50 and above
3. Male with symptomatic BPH.
4. IPSS symptom severity score ≥ 10
5. Peak urinary flow of < 12 ml/sec . Meeting the criterion on (2) two separate voiding trials , on a minimum voided volume of at least 125 cc for each voiding trial.
6. Prostate volume between 25 ml to 75 ml (assessed by ultrasound)
7. Blood CBC and biochemistry up to two weeks before screening demonstrating: Normal values of the PT, PTT and INR tests (anticoagulants should be stopped according to GCP)
8. Subject able to comply with the study protocol
9. Normal Urinalysis and urine culture

Exclusion Criteria:

1. Cardiac arrhythmias, cardiac disease including congestive heart failure, uncontrolled diabetes mellitus, significant respiratory disease, or known immunosuppression;
2. Neurogenic bladder and/or sphincter abnormalities due to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes
3. A post void residual (PVR) volume > 250 ml measured by ultrasound or acute urinary retention
4. Compromised renal function (i.e., serum creatinine level > 1.8 mg/dl, or upper tract disease);
5. Confirmed or suspected bladder cancer;
6. Recent (within 3 months) cystolithiasis or hematuria;
7. Urethral strictures, bladder neck contracture, urinary bladder stones or other potentially confounding bladder pathology;
8. An active urinary tract infection.
9. Enrolled in another treatment trial for any disease within the past 30 days.
10. Previous colo- rectal surgery (other than hemorrhoidectomy) or history of rectal disease if the therapy may potentially cause injury to sites of previous rectal surgery, e.g., if a transrectal probe is used;
11. Previous pelvic irradiation, cryosurgery or radical pelvic surgery;
12. Previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate
13. History of prostatitis within the past 5 years.
14. Median lobe obstruction of the prostate.
15. Cancer that is not considered cured, except basal cell or squamous cell carcinoma of the skin (cured defined as no evidence of cancer within the past 5 years).
16. Any serious medical condition likely to impede successful completion of the study
17. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.
18. Subjects who are actively taking medications that affects urination and BPH symptoms not completing the required washout period.
19. Baseline PSA ≥ 10 ng/ml.
20. Positive DRE.
21. Baseline PSA between 2.5-10 ng/ml and free PSA < 25%, without a subsequent negative prostate biopsy.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Pike, MD, Principal Investigator — St. John's Hospital
Locations (13):
- United States (11):
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Methodist Hospital, Brooklyn, New York
  - Winthrop University, Garden City, New York
  - St John's Episcopal, Lawrence, New York
  - Integrated Medical Professionals, Long Island City, New York
  - Manhattan Medical research, Manhattan, New York
  - Weill cornell, Manhattan, New York
  - Premier Urology Group, New York, New York
  - Primier Medical Center, Poughkeepsie, New York
  - Carolina Uro Research Center, Myrtle Beach, South Carolina
- Canada (2):
  - CIUSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - Toronto, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elterman D, Alshak MN, Martinez Diaz S, Shore N, Gittleman M, Motola J, Pike S, Hermann C, Terens W, Kohan A, Gonzalez R, Katz A, Schiff J, Goldfischer E, Grunberger I, Tu L, Kaminetsky J, Chughtai B. An Evaluation of Sexual Function in the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia in Men Treated with the Temporarily Implanted Nitinol Device. J Endourol. 2023 Jan;37(1):74-79. doi: 10.1089/end.2022.0226. Epub 2022 Oct 3. PMID 36070450
- See also: Company website — https://www.itind.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen centers participated in the study (14 in the United States, 2 in Canada) between July 2015 and October 2018.
  First patient was recruited on July 2015.
Pre-assignment Details: All patients on BPH related medications started a wash-out period prior to implantation: 1 month for alpha-blockers and 6 months for 5-alpha-reductase inhibitors (5-ARIs). Medication naïve patients seeking treatment refused medication in preference for a minimally invasive surgical technique.
Period: Overall Study
Arm/Group | iTind Arm | Sham Arm
Started | 128 | 57
Completed | 78 (78 patients reached 12 months FU visit.) | 57 (The Sham arm was analyzed up to 3 months FU visit as primary endpoint timeframe in accordance with the FDA guideline for BPH treatments, published in 2010, the most recent guidance available at the time of the study.)
Not Completed | 50 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iTind Arm | Sham Arm | Total
Number analyzed (Participants) | 128 | 57 | 185
Age, Customized [Mean (Standard Deviation); unit: years] | 61.5 (6.5) | 60.1 (6.3) | 61.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 128 | 57 | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 23 | 11 | 34
  White | 86 | 36 | 122
  More than one race | 16 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
IPSS score [Mean (Standard Deviation); unit: units on a scale] — The International Prostate Symptom Score. Scale: minimum 0 (zero), maximum 35. Lower values are better.
  units on a scale | 22.1 (6.8) | 22.8 (6.2) | 22.3 (6.6)
Qmax [Mean (Standard Deviation); unit: ml/sec] | 8.7 (3.3) | 8.5 (2.4) | 8.6 (3.0)
PVR [Mean (Standard Deviation); unit: ml] — Post-Void Residual is the amount of urine left in the bladder at the end of micturition.
  PVR varies in a given individual and is measured in ml. Lower values are better.
  ml | 61.6 (55.5) | 61.9 (54.2) | 61.6 (55.0)
QoL [Mean (Standard Deviation); unit: units on a scale] — Quality of Life Scale: minimum 0 (zero), maximum 5. Lower values are better.
  units on a scale | 4.6 (1.3) | 4.9 (1.0) | 4.6 (1.2)
IIEF questionnaire [Mean (Standard Deviation); unit: units on a scale] — The International Index of Erectile Function score. Scale: minimum 6, maximum 75. Higher values are better.
  units on a scale | 38.3 (20.7) | 39.1 (19.6) | 38.5 (20.3)
SHIM questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Sexual Health Inventory for Men questionnaire. Scale: minimum 1, maximum 25. Higher values are better.
  units on a scale | 13.2 (7.3) | 14.2 (6.6) | 13.5 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Month 3 Results in the IPSS Score in Both Arms.
Description: Month 3 results in the IPSS Score in both arms IPSS - The International Prostate Symptom Score. Scale: minimum 0 (zero), maximum 35. Lower values are better.
Time Frame: 3 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | iTind Arm | Sham Arm
Number analyzed (Participants) | 128 | 57
score on a scale | 12.57 (6.95) | 15.8 (9.0)

2. Secondary Outcome: Qmax Measurement
Description: Month 3 results in Qmax (maximum urinary flow rate)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | iTind Arm | Sham Arm
Number analyzed (Participants) | 128 | 57
ml/sec | 13.55 (6.4) | 11.4 (5.3)

3. Secondary Outcome: PVR
Description: Month 3 results in PVR (post-void residual urine volume)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | iTind Arm | Sham Arm
Number analyzed (Participants) | 128 | 57
ml | 59.44 (56.43) | 66.9 (65.1)

4. Secondary Outcome: IIEF Questionnaire
Description: The International Index of Erectile Function score. Scale: minimum 6, maximum 75. Higher values are better. Month 3 results in IIEF.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTind Arm | Sham Arm
Number analyzed (Participants) | 128 | 57
score on a scale | 43.52 (22.24) | 40.5 (22.8)

5. Secondary Outcome: SHIM
Description: The Sexual Health Inventory for Men questionnaire. Scale: minimum 1, maximum 25. Higher values are better. Month 3 results in SHIM.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTind Arm | Sham Arm
Number analyzed (Participants) | 128 | 57
score on a scale | 13.7 (7.76) | 13.2 (7.9)

ADVERSE EVENTS:
Time Frame: Adverse Events were documented from implantation day until the first follow up visit at 3 months.
Description: AEs and SAEs defined in the same manner as clinicaltrials.gov.
Groups:
- iTind Arm: iTind implant is implant during the study for 5-7 days. Temporary Implantable Nitinol Device (iTIND).
- Sham Arm: Foley catheter is used during the study. Foley catheter will be placed and immediately removed.
Arm/Group | iTind Arm | Sham Arm
All-Cause Mortality (participants affected / at risk) | 1/128 | 0/57
Serious Adverse Events (participants affected / at risk) | 10/128 | 2/57
Other Adverse Events (participants affected / at risk) | 45/128 | 5/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTind Arm (N=128) | Sham Arm (N=57)
Urinary retention (Renal and urinary disorders) | 2 (16) | 0 (0) — One case Injury relates to poisoning and procedural complications and the second one relates to renal and urinary disorders
Urinary tract infection (Infections and infestations) | 2 (16) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (16) | 0 (0)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (16) | 0 (0) — One patient died from an unrelated pancreatic cancer complication.
General weakness (General disorders) | 2 (16) | 0 (0) — General system disorders NEC
Nausea and vomiting (Gastrointestinal disorders) | 2 (16) | 0 (0) — Nausea and vomiting symptoms
Depression, suicidal and self-injurious behavior (Psychiatric disorders) | 2 (16) | 0 (0)
Abscess and sepsis (Infections and infestations) | 2 (16) | 0 (0)
Deep vein thrombosis (DVT) of legs (Vascular disorders) | 1 (16) | 0 (0) — Peripheral embolism and thrombosis
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (16) | 0 (0) — Upper limb fractures and dislocations
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Central nervous system vascular disorders (Nervous system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTind Arm (N=128) | Sham Arm (N=57)
Dysuria (Renal and urinary disorders) | 27 (109) | 5 (19)
Hematuria (Renal and urinary disorders) | 16 (109) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (109) | 0 (0)

LIMITATIONS AND CAVEATS:
Since the study included specific inclusion criteria in regards to age, IPSS, Qmax and prostate volume, our results are not generalizable to all men with LUTS secondary to BPH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02506465/Prot_SAP_000.pdf